CLINICAL TRIAL: NCT05932680
Title: Phase 2, Single-Arm, Non-Inferiority Study Of Limited-Duration Teclistamab For Relapsed Refractory Multiple Myeloma
Brief Title: Limited-duration Teclistamab
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UPCC 08423; IRB 853459 (Other: University of Pennsylvania)
Record Dates: First submitted 2023-06-08; First posted 2023-07-06 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Myeloma Multiple
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Teclistamab is the study drug. The intervention is the cessation of the drug.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Off Drug Surveillance (Experimental): Participants will stop receiving teclistamab and will be monitored closely for growth of their multiple myeloma. Participants will restart teclistamab if their multiple myeloma starts to grow.
  Interventions: Other: Off Drug Surveillance

INTERVENTIONS:
Other: Off Drug Surveillance — After stopping teclistamab, participants will be monitored monthly by standard serum paraprotein studies for disease progression. Participants will resume teclistamab at time of disease progression. After Teclistamab therapy re-initiation on-study, monthly response assessments and data for other study endpoints will be obtained. All participants will undergo peripheral blood collection for correlative research studies at baseline and every two months on-study. Participants who enroll on the biomarker sub-study will undergo bone marrow examination and peripheral blood collection for correlative studies at study entry, at time of disease progression and at six months from enrollment.

SUMMARY:
This is a single-arm, non-inferiority study in which patients who have achieved a very good partial response (VGPR) or better, according to International Myeloma Working Group (IMWG) response criteria, following 6 to 9 months of treatment with teclistamab, a B-cell maturation antigen (BCMA)-directed T-cell engager (anti-BCMAxCD3 bispecific antibody), will be offered monitored drug discontinuation. Teclistamab is typically dosed on a regular schedule (every 1-4 weeks) indefinitely until disease progression ("continuous therapy"). Here, a limited-duration regimen will be studied in which patients achieving ≥VGPR after 6-9 months of standard teclistamab dosing will discontinue therapy and resume if laboratory or clinical parameters suggest early disease progression ("limited-duration therapy"). Patients will enter the clinical trial protocol after completing 6-9 months of standard teclistamab monotherapy and achieving ≥VGPR. The study's hypothesis is that the failure probability six months after stopping teclistamab in this patient population will be non-inferior compared to that of historical controls treated with continuous therapy. Reducing drug exposure may be beneficial by reducing risk of infection and reducing anti-BCMA selective pressure toward generation of BCMA-negative relapses. Analysis of minimal residual disease (MRD), tumor features, and bone marrow microenvironment parameters, which will be pursued as exploratory correlative analyses in this study, may identify factors that predict durable response to limited-duration therapy and thereby enable more precise selection of patients likely to benefit from this approach. A subset of patients will be enrolled on a biomarker study for analysis of these exploratory endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be age ≥18 and able to give written, informed consent.
* Participants must have initiated teclistamab (first full dose) 6-9 months prior to enrollment and received an average teclistamab dose of at least 1.5 mg/kg/month since the date of the first 1.5 mg/kg dose.
* Participants must have received a teclistamab dose within 4 weeks prior to enrollment.
* Participants must have had measurable disease according to IMWG criteria within 1 month prior to teclistamab initiation or first full teclistamab dose
* Participants must have achieved a confirmed VGPR or better to teclistamab therapy at any assessment prior to enrollment and have ongoing response (i.e., no disease progression) at time of enrollment per IMWG consensus criteria (Appendix 14.3).
* Prior to initiating teclistamab, participants must have received therapy with a proteasome inhibitor, thalidomide analog (lenalidomide or pomalidomide), and an anti-CD38 antibody and meet one of the following criteria:

  1. ≥3 prior lines of therapy (with lines-of-therapy delineated according to IWMG guidelines)
  2. Refractory to both a proteasome inhibitor and a thalidomide analog.
* Participants must have had an ECOG performance status of 0-2 at time of teclistamab initiation; in addition, ECOG performance status must be 0-1 at time of enrollment.
* Participants must not have known diagnoses of systemic amyloidosis or POEMS syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Failure free at six months following teclistamab discontinuation | Six months after teclistamab discontinuation
  Failure-free survival is defined as the rate of evaluable individuals who have not experienced any of the following predefined failure events within 6 months of discontinuing teclistamab. Failure is defined as earliest occurrence of any of the following: Participants who progress by IMWG criteria after discontinuing teclistamab, failure to achieve at least minimal response within 90 days after reinitiating teclistamab or failure to resume teclistamab within 90 days of IMWG-defined disease progression. Participants who reinitiate teclistamab due to rise in disease markers before IMWG criteria for disease progression are met, disease progression by IMWG criteria after reinitiation of teclistamab. Initiation of non-teclistamab systemic multiple myeloma therapy. Failure date will be defined as the date of initiating subsequent therapy. Death due to complications of multiple myeloma, teclistamab therapy, or infection

SECONDARY OUTCOMES:
Time to progression and progression-free survival | Two years after teclistamab discontinuation.
  Time-to-progression and progression-free survival by IMWG criteria from time of teclistamab discontinuation, using the best response to initial teclistamab course as the baseline for scoring disease progression.
Time-to-treatment failure | Two years after teclistamab discontinuation
  Time-to-treatment failure as defined in the primary endpoint
Re-initiation rate | Six months after teclistamab discontinuation
  Proportion of subjects who re-initiate teclistamab within six months following discontinuation
Rate of response to teclistamab re-initiation | Two years after teclistamab discontinuation
  Among subjects with IMWG-defined measurable disease at time of teclistamab re-initiation, overall response rate (PR or better) and clinical benefit rate (minimal response or better) to teclistamab upon re-initiating therapy.
Rate of infectious complications | 12 months after teclistamab discontinuation
  Frequency of infectious complications from time of teclistamab discontinuation.
Rate and type of clinical complications of progressive disease | Six months after teclistamab discontinuation
  Frequency of the type and rate of clinical complications of progressive disease (e.g., new osteolytic lesions) from time of teclistamab discontinuation through 6 months post-discontinuation.
Quality of life | Two years after teclistamab discontinuation
  QOL is measured using the MM-FACT instrument. Health-related quality of life (HRQoL) as measured by Functional Assessment of Cancer Therapy - Multiple Myeloma (FACT-MM) questionnaire score at enrollment and monthly post-enrollment assessments. The higher the score, the better the quality of life. Two scores will be derived - FACT-MM Trial Outcome Index (TOI) (range: 0-112) and FACT-MM total score (range: 0-164).
Mean percent change in peripheral blood studies | Two years after teclistamab discontinuation
  Mean percent change in peripheral blood cell counts, immunoglobulin levels, and T cell counts (total and CD4/CD8 subsets) from the time of enrollment through teclistamab resumption and through the end-of-study.

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Garfall, MD, Principal Investigator — Penn Medicine
Locations (5):
- United States (5):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Columbia University, New York, New York
  - Abramson Cancer Center at University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Honickman Center, Philadelphia, Pennsylvania